CLINICAL TRIAL: NCT06509672
Title: Combined Effects of Plyometric and Endurance Training on Speed, Agility and Strength Among Female Hockey Players
Brief Title: Combined Effects of Plyometric and Endurance Training Among Female Hockey Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0469
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Plyometric Exercise; Endurance Training; Hockey
Keywords: Plyometric training; Endurance training; Hockey players
MeSH Terms: interventions — Endurance Training; Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Plyometric and Endurance Training (Experimental): will receive both below mentioned trainings with alternative timings
  Interventions: Other: Combined Plyometric and Endurance Training
- Plyometric Training (Active Comparator): First of all, the training session will be started with a warm-up period of 10min. the athlete will be asked to do gentle warm-up exercises. In the next step of training Counter movement jump for Plyometric training (CMJ will be performed with a squat starting position, that is, knees flexed to 90 ° and hands on hips. From this position, the hockey players will be required to bend their knees to a freely chosen angle and perform a maximal vertical thrust. The hands are held on the hips during the jump to avoid any effect of arm-swinging. Participants will be instructed to keep their body vertical throughout the jump, avoiding undue lateral and frontal movements, and to land with knees fully extended.) The CMJ period will be in 2 rounds each round of 8 min with 4 min break between the rounds. The training session will end with a 10min cooling period. The complete plyometric training session will be of 40mins.
  Interventions: Other: Plyometric Training
- Endurance Training (Active Comparator): Endurance training will be done on a cycle ergometer. Subjects will initially do six 3-min bouts of exercise with 3-min rest periods between bouts. The bouts will be done at power outputs corresponding to that which require 60 and 80% VO₂ max respectively. After 4 weeks a seventh bout will be added and after 8 weeks an eight bout. After 10 weeks 10 bouts will be done till the end of the training. Each endurance training sub-session will last for 35-45 min.
  Interventions: Other: Endurance training

INTERVENTIONS:
Other: Combined Plyometric and Endurance Training — this include Combined Plyometric and Endurance Training for 12 weeks
  Arms: Combined Plyometric and Endurance Training
Other: Plyometric Training — this include Plyometric Training for 12 weeks
  Arms: Plyometric Training
Other: Endurance training — this include Endurance Training for 12 weeks
  Arms: Endurance Training

SUMMARY:
Athletes need plyometric training as well as endurance training to enhance their speed, strength and agility in the field. Plyometric exercise involves stretching the muscle immediately before making a rapid concentric contraction. The combined action is commonly called a stretch-shortening cycle (SSC). Similar gains of maximal strength have been reported with traditional strength and plyometric training, but the latter approach appears to induce greater gains in muscle power. The combination of balance and muscle strength/power exercises seems to be an appropriate possibility, since both modalities induced adaptation on the neuromuscular level. A blocked combination of balance and muscle strength exercises effectively improve physical performance, and improvements in performance are more pronounced if balance exercises are followed by strength exercises than vice versa.

DETAILED DESCRIPTION:
Strength and endurance training are often done concurrently by fitness enthusiasts and athletes. Concurrent strength and endurance training however, result in "antagonism" of the training responses. Combined strength and endurance training in previously untrained subjects has developed strength impairment in comparison to strength training alone, whereas endurance development, expressed as increases in maximal aerobic power has not been impaired. A combination of some forms of strength and endurance training maybe "addictive" rather than antagonistic. Some endurance training programs have increases strength and muscle fiber size. A randomized controlled trial will be conducted. Non-probability convenient sampling technique will be used. Study will be carried in hockey clubs at Lahore. Only female players of age 18-24 with one year experience in hockey, only players who will participate in all training sessions will be included in the statistical analysis. Participants with the history of systemic disease, with history of lower extremity and lumber spine pathology, with prior surgery history and participants having injuries resulting in loss of one or more hockey matches/ training sessions in the preceding three months prior to the initiation of the study will be excluded. Three groups will be included in the study each containing 10 participants. Group A will be given plyometric training for 12 weeks, Group B will be given endurance training for 12 weeks and Group C will be given both trainings for 12 weeks. Pre-training values will be taken prior training. Mid-training values will be taken after 6 weeks of training and post-training values will be taken after training.

ELIGIBILITY:
Inclusion Criteria:

* Only female hockey players

  * Age 18-24 years
  * Athletes with at least one year experience in hockey
  * Athletes must be without previous experience in intense strength/endurance training
  * Only players who will participate in at all training sessions will be included in the statistical analysis

Exclusion Criteria:

* Participants having injuries resulting in loss of one or more hockey matches/ training sessions in the preceding three months prior to the initiation of the study
* Participants with the history of systemic disease
* Participants with history of lower extremity and lumber spine pathology
* Participants with prior surgery history

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
Speed | 0 week, 6 week, 12 week
  will be measured by Sprint test
Agility | 0 week, 6 week, 12 week
  will be measured by t test
Strength | 0 week, 6 week, 12 week
  will be measured by 5 jump distance test

CONTACTS AND LOCATIONS:
Overall Officials: Awishbah Khan, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Academy, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chelly MS, Ghenem MA, Abid K, Hermassi S, Tabka Z, Shephard RJ. Effects of in-season short-term plyometric training program on leg power, jump- and sprint performance of soccer players. J Strength Cond Res. 2010 Oct;24(10):2670-6. doi: 10.1519/JSC.0b013e3181e2728f. PMID 20844458
- [Background] Sale DG, Jacobs I, MacDougall JD, Garner S. Comparison of two regimens of concurrent strength and endurance training. Med Sci Sports Exerc. 1990 Jun;22(3):348-56. PMID 2381303
- [Background] Muehlbauer T, Wagner V, Brueckner D, Schedler S, Schwiertz G, Kiss R, Hagen M. Effects of a blocked versus an alternated sequence of balance and plyometric training on physical performance in youth soccer players. BMC Sports Sci Med Rehabil. 2019 Sep 2;11:18. doi: 10.1186/s13102-019-0131-y. eCollection 2019. PMID 31497301
- [Background] Markov A, Hauser L, Chaabene H. Effects of Concurrent Strength and Endurance Training on Measures of Physical Fitness in Healthy Middle-Aged and Older Adults: A Systematic Review with Meta-Analysis. Sports Med. 2023 Feb;53(2):437-455. doi: 10.1007/s40279-022-01764-2. Epub 2022 Oct 12. PMID 36222981
- [Background] Aloui G, Souhail H, Hayes LD, Bouhafs EG, Chelly MS, Schwesig R. Effects of Combined Plyometric and Short Sprints Training on Athletic Performance of Male U19 Soccer Players. Front Psychol. 2021 Sep 15;12:714016. doi: 10.3389/fpsyg.2021.714016. eCollection 2021. PMID 34603139